CLINICAL TRIAL: NCT04505943
Title: Comparison of Vaginal Misoprostol and Dinoprostone and Isonicotinic Acid Hydrazide Prior to Copper Intrauterine Device Insertion in Nulliparous Women : a Randomized Controlled Study
Brief Title: Vaginal Misoprostol and Dinoprostone and Isonicotinic Acid Hydrazide Prior to Copper Intrauterine Device Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/352/5/19
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: IUCD Complication
MeSH Terms: interventions — Isoniazid; KLK15 protein, human; Misoprostol

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- isonicotinic acid hydrazide (Experimental): 2vaginal tablet of isonicotinic acid hydrazide inserted by the study nurse12 hours before IUD insertion.
  Interventions: Drug: Isonicotinic Acid Hydrazide
- dinoprostone (Active Comparator): 2 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 12 hours before IUD insertion.
  Interventions: Drug: dinoprostine
- misoprostol (Active Comparator): 2 vaginal tablet of misoprostol (200 mcg) (Misotac®; Sigma Pharma, SAE, Egypt) inserted by the study nurse 12hours before IUD insertion.
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: Isonicotinic Acid Hydrazide — 2 vaginal tablet of isonicotinic acid hydrazide inserted by the study nurse12 hours before IUD insertion.
  Other Names: INH
  Arms: isonicotinic acid hydrazide
Drug: dinoprostine — 2 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 3 hours before IUD insertion.
  Other Names: prostin
  Arms: dinoprostone
Drug: misoprostol — 2 vaginal tablet of misoprostol (200 mcg) (Misotac®; Sigma Pharma, SAE, Egypt) inserted by the study nurse 3 hours before IUD insertion
  Other Names: Misotac
  Arms: misoprostol

SUMMARY:
To compare the effect of vaginal dinoprostone versus vaginal misoprostol and Isonicotinic Acid Hydrazide administered before the copper intrauterine device(IUD) insertion in reducing IUD inertion pain and the difficulty in inserting the IUD in nulliparous women.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women requesting copper IUD insertion

Exclusion Criteria:

* pregnancy,
* Parous women,
* contraindications or allergy to dinoprostone or misoprostol,contraindication to IUD insertion,
* untreated active cervicitis or vaginitis,
* undiagnosed abnormal uterine bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — nulliparous women
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The difference in visual analog scale pain scores during intrauterine device insertion | 10 minuts
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

SECONDARY OUTCOMES:
the difference in visual analog scale pain scores during tenaculum application | 10 minuts
  The difference in pain scores during tenaculum application using a visual analog scale from 0 to 10
the ease of IUD insertion | 10 minutes
  the ease of IUD insertion using ease of insertion score from 0 to 10 cm (0 = very easy insertion, 10 cm = terribly difficult insertion)
women's satisfaction level: score | 10 minutes
  women's satisfaction level using satisfaction score from 0 to 10 cm where 0 denotes no satisfaction and 10 denotes maximum satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No